CLINICAL TRIAL: NCT01509469
Title: The Effect of Different Macronutrients on Ileal Brake Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Principal Investigator, Mark van Avesaat, MD, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NL36916.068.11
Record Dates: First submitted 2011-08-09; First posted 2012-01-13 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Obesity; Overweight
Keywords: Ileal brake; Casein; Sucrose; Ileal infusion
MeSH Terms: conditions — Obesity; Overweight | interventions — Caseins; Sucrose; Sodium Chloride; Safflower Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Low dose casein (Experimental): Ileal infusion of low dose casein
  Interventions: Dietary Supplement: Casein
- High dose casein (Experimental): Ileal infusion of high dose casein
  Interventions: Dietary Supplement: Casein
- Low dose sucrose (Experimental): Ileal infusion of low dose sucrose
  Interventions: Dietary Supplement: Sucrose
- High dose sucrose (Experimental): Ileal infusion of high dose sucrose
  Interventions: Dietary Supplement: Sucrose
- Placebo (Placebo Comparator): Ileal infusion saline
  Interventions: Other: Saline
- Safflower oil (Active Comparator): Ileal infusion safflower oil
  Interventions: Dietary Supplement: Safflower oil

INTERVENTIONS:
Dietary Supplement: Casein — Ileal infusion of low dose casein (5 gram)
  Arms: Low dose casein
Dietary Supplement: Casein — Ileal infusion of high dose casein (15 gram)
  Arms: High dose casein
Dietary Supplement: Sucrose — Ileal infusion of low dose sucrose (4.3 gram)
  Arms: Low dose sucrose
Dietary Supplement: Sucrose — Ileal infusion of high dose sucrose (12.9 gram)
  Arms: High dose sucrose
Other: Saline — Ileal infusion with saline (180mL in total)
  Arms: Placebo
Dietary Supplement: Safflower oil — Ileal infusion with safflower oil (6gr safflower oil in water)
  Arms: Safflower oil

SUMMARY:
The purpose of this study is to determine whether ileal infusion of casein and sucrose can activate the ileal brake.

DETAILED DESCRIPTION:
The appearance of a food matrix into the duodenum, both during a meal and during the postprandial phase results in a feed-back from different parts of the intestine to the stomach, to the small intestine and to the central nervous system. All these processes inhibit, in concert, food processing in the gastrointestinal tract, satiation and appetite sensations and, consequently, food intake. These processes are involved in the so-called intestinal brake. The location at which the feedback process is initiated determines the severity of the brake effect; the entry of nutrients into the duodenum and jejunum activates the so-called duodenal and jejunal "brakes": negative feedback mechanisms that influence the function of more proximal parts of the gastrointestinal tract. Activation of both of these feedback mechanisms results in reduction of food intake and inhibition of hunger, probably partly by inhibition of gastric emptying rate (thus contributing to enhanced and prolonged gastric distension) and small intestinal transit time. More distal in the small intestine, the ileal brake is a feedback mechanism that results in inhibition of proximal gastrointestinal motility and secretion and increase feelings of satiation and reduction of ad libitum food intake.These results all point to a potentially powerful role of the ileal brake in the regulation of digestion, with direct or indirect impact upon eating behaviour and satiation.

The current scientific data strongly suggest that activation of the ileal brake provides the most powerful feedback mechanism to gastrointestinal transit and, especially, satiety signals and food intake. Most studies have used fat as macronutrient. The effects of several amounts, types and preparations of fat on the ileal brake have previously been investigated and reported.

Until present, the effects of the other macronutrients to induce the ileal brake remain largely unknown. There is evidence that carbohydrates induce the ileal brake. Proteins may also exert effects, although data are scarce and not convincing. However, it becomes more and more accepted that proteins may induce stronger effects on satiation and food intake than fat or carbohydrates.

In this study we're going to investigate the effect of intraileal infusion of casein and sucrose on ileal brake activation.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history and previous examination, no gastrointestinal complaints can be defined.
* Age between 18 and 55 years. This study will include healthy adult subjects (Male and Female), Women must be taking oral contraceptives. Subjects over 55 years have an increased risk for comorbidities, therefore, subjects over 55 years will not be included.
* BMI between 18 and 29 kg/m2
* Less then 2 'yes' responses in the SCOFF questionnaire (see appendix F1)
* Weight stable over at least the last 6 months

Exclusion Criteria:

* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol. The severity of the disease (major interference with the execution of the experiment or potential influence on the study outcomes) will be decided by the principal investigator.
* Use of medication, including vitamin supplementation, except oral contraceptives, within 14 days prior to testing
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study
* Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgement of the principle investigator)
* Dieting (medically prescribed, vegetarian, diabetic, macrobiological, biological dynamic)
* Pregnancy, lactation
* Excessive alcohol consumption (>20 alcoholic consumptions per week)
* Smoking
* Blood donation within 3 months before the study period
* Self-admitted HIV-positive state
* Eating disorders detected using the 'SCOFF questionnaire' (in Dutch translation)
* Lactose or cow milk intolerance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Difference in satiation (as measured by VAS) and food intake as measured during an ad libitum meal | 1 day

SECONDARY OUTCOMES:
Measurements in plasma and/or platelet poor plasma Plasma levels of the gut hormone Cholecystokinin (CCK) | 1 day
Gastric emptying by using the C13 stable isotope breath test | 1 day
Small bowel transit time by using lactulose hydrogen breath test | 1 day
Gallbladder volumes by gallbladder ultrasound | 1 day
Measurements in plasma and/or platelet poor plasma Plasma levels of the gut hormone Glucagon Like Peptide-1 (GLP-1) | 1 day
Measurements in plasma and/or platelet poor plasma Plasma levels of the gut hormone peptide YY (PYY) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: A. Masclee, Prof., Principal Investigator — Maastricht University Medical Centre +
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Ripken D, van Avesaat M, Troost FJ, Masclee AA, Witkamp RF, Hendriks HF. Intraileal casein infusion increases plasma concentrations of amino acids in humans: A randomized cross over trial. Clin Nutr. 2017 Feb;36(1):143-149. doi: 10.1016/j.clnu.2016.01.012. Epub 2016 Jan 29. PMID 26872548